CLINICAL TRIAL: NCT02571426
Title: The Influence of Propofol and Sevoflurane Anesthesia on Water and Sodium Retention in Children
Brief Title: Renal Function During Pediatric Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Micael Taavo, Staff physician, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SRC52320142569-1
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Renal Failure; Anesthesia
MeSH Terms: conditions — Renal Insufficiency | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Continuous infusion during surgery. Individual dosage.
  Interventions: Drug: propofol
- sevoflurane (Active Comparator): Inhalational anesthetic during surgery. Individual dosage
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — anesthetic agent
  Other Names: sevorane
  Arms: sevoflurane
Drug: propofol — anesthetic agent
  Other Names: diprivane
  Arms: Propofol

SUMMARY:
It is known that volatile anesthesia, such as sevoflurane, retain water and that this appears more pronounced in children. However, the mechanisms for this effect is unknown and it is not clear if the commonly used anesthetic propofol does the same. In this study the investigators want to compare the fluid and electrolyte conserving effects of sevoflurane and propofol in a pediatric setting and also investigate humoral changes induced by these anesthetics.

DETAILED DESCRIPTION:
Prior studies by the investigators research group have shown water and sodium retention in experimental animals undergoing sevoflurane anesthesia. Preliminary data suggest that this is not as obvious with propofol anesthesia. The investigators aim to study if this difference is present in children.

Subjects are collected from ordinary routine operations of hypospadia. By routine, all boys undergoing this surgery get a sacral blockade and a urine catheter. The children are randomized to either sevoflurane or propofol anesthesia. Before or immediately after induction of anesthesia baseline blood samples are collected for analysis of sodium, potassium, creatinine, osmolality, angiotensin II, arginine-vasopressin and aldosterone. Perioperative fluids are started, a balanced glucose infusion with 132mmol sodium content, covering basal fluid need + 20%. This infusion is continued until the end of the protocol at the ward. At the induction of anesthesia the investigators start measuring urine output every 20th minute. The same blood samples as above are collected again during mid-operation. At the end of anesthesia the investigators collect all the urine and send a sample for urine analysis of sodium, potassium, osmolality and creatinine.

In the postoperative ward the investigators again start collecting urine every 20 minutes for 120 minutes. All urine after 120 minutes are collected, and a sample sent for analysis. After 60 minutes at the postoperative ward, blood samples are again collected for analysis.

In the childrens ward the protocol for the postoperative ward is repeated, with urine collection and sample, as well as blood samples. After 120 minutes the protocol ends.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for hypospadia surgery.

Exclusion Criteria:

* American Association of Anesthesiology class above 2
* Weight above 50 kg or below 10 kg
* Hypersensitivity towards the anesthetic agents (difficult peanut or soy allergy)
* Inability for parent to understand study information

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2018-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
urine output during anesthesia | 2 hours

SECONDARY OUTCOMES:
urine output postoperatively | 4 hours
sodium excretion postoperatively | 4 hours
Changes in aldosterone, angiotensin II, arginine-vasopressin during surgery | 2 hours
  Comparison of blood samples of fluid balance regulatory hormones collected at baseline, during surgery and 1 hour + 3 hours postoperatively
Changes in aldosterone, angiotensin II, arginine-vasopressin postoperatively | 4 hours
  Comparison of blood samples of fluid balance regulatory hormones collected at baseline, during surgery and 1 hour + 3 hours postoperatively
Sodium excretion during anesthesia | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Micael Taavo, MD, Principal Investigator — Uppsala University
Locations (1):
- Akademiska university hospital, Uppsala, Sweden